CLINICAL TRIAL: NCT05507203
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase III Study to Evaluate the Efficacy and Safety of ABX464 Once Daily for Induction Treatment in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: ABTECT-1 - ABX464 Treatment Evaluation for Ulcerative Colitis Therapy -1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABX464-105
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ABX464

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ABX464 50mg (Experimental): Subjects will be orally dosed daily in a fed condition ideally at the same time in the morning) for 8 weeks
  Interventions: Drug: ABX464
- ABX464 25mg (Experimental): Subjects will be orally dosed daily in a fed condition ideally at the same time in the morning) for 8 weeks
  Interventions: Drug: ABX464
- Placebo (Placebo Comparator): Subjects will be orally dosed daily in a fed condition ideally at the same time in the morning) for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABX464 — Administered once daily in the morning with food
  Other Names: Obefazimod
  Arms: ABX464 25mg; ABX464 50mg
Drug: Placebo — Administered once daily in the morning with food
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, placebo controlled study to evaluate the efficacy and safety of ABX464 given at 25 or 50 mg QD in inducing clinical remission in subjects with moderately to severely active ulcerative colitis who have inadequate response, no response, a loss of response, or an intolerance to either conventional therapies [corticosteroids, immunosuppressant (i.e. azathioprine, 6-mercaptopurine, methotrexate)] and/or advanced therapies [biologics (TNF inhibitors, anti-integrins, anti-IL-23), and/or S1P receptor modulators, and/or JAK inhibitors].

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 16 years old; Adolescent subjects will only be enrolled if approved by the country regulatory/health authority. If these approvals have not been granted, only subjects ≥ 18 years old will be enrolled. To be eligible, adolescent subjects must weight ≥ 40 kg and meet the definition of Tanner Stage 5 at the screening visit.
* Subjects must understand, sign and date the written voluntary informed consent form at the visit prior to any protocol-specific procedures. For under-aged subjects, national requirements regarding consent should also be met.
* Documented diagnosis of UC confirmed by endoscopy and histology. Should endoscopy/histology results not be available at screening, results from endoscopies or biopsies taken at screening may be used.
* Active disease defined by modified Mayo score (MMS) ≥ 5 with rectal bleeding subscore (RBS) ≥ 1 and endoscopy subscore (MES) of 2 or 3 (confirmed by central reader).
* Subjects with documented inadequate response (defined as lack of response or loss of response or intolerance) to at least one of the following treatments: corticosteroids, immunosuppressant, biologic or biosimilar therapies, S1P receptor modulators and/or JAK inhibitors and/or new drugs approved during the study (note: failure to only 5-ASA or sulfasalazine is not accepted).
* Women of childbearing potential (WOCBP) subjects and male subjects with WOCBP partner must agree to comply with the contraception requirements described in the protocol.
* Subjects able and willing to comply with study visits and procedures as per protocol.
* Subjects should be affiliated to a health insurance policy whenever required by a participating country or state.

Exclusion Criteria:

* Subjects with UC limited to an isolated proctitis (≤ 15cm from anal verge) determined by endoscopy central reading.
* Subjects with primary sclerosing cholangitis or autoimmune hepatitis.
* Subjects who have failed on 5-ASA or sulfasalazine therapy only.
* Subjects with CD or presence or history of fistula, indeterminate colitis, infectious/ischemic colitis or microscopic colitis (lymphocytic and collagenous colitis).
* History or current evidence of toxic megacolon, fulminant colitis, bowel perforation.
* History of colonic cancer or colonic low grade or high grade dysplasia adenomatous polyps, and/or at the screening endoscopy, evidence of colonic cancer or evidence of low grade or high grade dysplasia adenomatous polyps (fully removed or not).
* Recent or planned bowel surgery or history of proctocolectomy or partial colectomy or current stoma.
* Subjects on antidiarrheals including those working on motility (e.g., loperamide, diphenoxylate with atropine, etc.).
* Subjects on probiotics (e.g., Culturelle® [Lactobacillus GG, i-Health, Inc.], Saccharomyces boulardii).
* Subjects who do not meet the washout period requirements prior to the screening endoscopy
* Subjects with the following hematological and biochemical laboratory parameters obtained during the screening period:

  * Hemoglobin ≤ 8.0 g dL-1
  * Absolute neutrophil count < 750 mm-3
  * Platelets < 100,000 mm-3
  * Creatinine clearance < 60 mL.min-1 (Cockroft-Gault formula)
  * Total serum bilirubin > 1.5 x ULN
  * Alkaline phosphatase, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2 x ULN
* Subjects with the following conditions (infection):

  * Subjects with chronic or recurrent grade 3 or grade 4 infection within the last 2 months prior to screening or a history of opportunistic infection while not on immunosuppressive therapy.
  * Herpes zoster reactivation within the last 2 months prior to screening.
  * Subjects with active infection at screening or any major episode of infection that required hospitalization or treatment with intravenous antibiotics within 1 month of screening or during screening. Fungal infection of nail beds is allowed.
  * Positive assay or stool culture for pathogens (ova and parasite examination, bacteria) or positive test for Clostridium difficile toxin at screening. If C. difficile is positive, subject may be treated and retested ≥ 2 weeks after completing treatment.
  * Subjects with HIV infection.
  * Subjects having acute or chronic hepatitis B infection at screening (positive for hepatitis B surface antigen [HbsAg], or negative for HbsAg and positive for anti-hepatitis B core antibody in conjunction with detectable HBV DNA, or detectable HBV DNA).
  * Subjects having acute or chronic hepatitis C infection at screening as defined by positive for hepatitis C antibody (subjects successfully treated and without recurrence ≥ 1 year with no detectable HCV RNA [assessed centrally] are eligible).
  * Active tuberculosis (TB) or untreated latent TB are ruled out. For subjects with positive or intermediate QuantiFERON test see study protocol.
* Subjects with an uncontrolled ischemic heart disease and/or a history of congestive heart failure with New York Heart Association (NYHA) class 3 or 4 symptoms.
* Subjects with a family or personal history of congenital or acquired long QT syndrome, or subjects with a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval [Fridericia or Bazett correction] >450 milliseconds for male and > 460 milliseconds for female).
* Subjects with a history of torsade de pointe (TdP).
* Acute or chronic of clinically relevant pulmonary, hepatic, pancreatic or renal functional abnormality, encephalopathy, neuropathy or unstable central nervous system pathology such as seizure disorder, or any other clinically significant medical problems as determined by physical examination and/or laboratory screening tests and/or medical history (note: treated autoimmune hypothyroidy and autoimmune diabetes are allowed).
* Serious illness requiring hospitalization within 4 weeks prior to screening (except UC flare).
* Subjects previously treated with ABX464.
* Subjects with a known hypersensitivity to the active substance or to any of the excipients.
* WOCBP subject who is pregnant or breast-feeding at screening, or intends to become pregnant during the study, or male subject with WOCBP partner who intends to be pregnant during the study.
* Illicit drug or alcohol abuse or dependence.
* Subjects who received live vaccine within 3 months prior to screening and/or who's planning to receive such a vaccine during the study duration.
* Use of any investigational or non-registered product within 3 months or within 5 half-lives preceding baseline, whichever is longer, and during the study.
* Subjects committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.
* Any condition, which in the opinion of the investigator, could compromise the subject's safety or adherence to the study protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 639 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve clinical remission per Modified Mayo Score at week 8 | 8 weeks
  To compare the efficacy of ABX464 versus placebo on clinical remission

SECONDARY OUTCOMES:
Proportion of subjects who achieve endoscopic improvement at week 8 | 8 weeks
  To compare the efficacy of ABX464 versus placebo on endoscopic improvement
Proportion of subjects who achieve clinical response per MMS at week 8 | 8 weeks
  To compare the efficacy of ABX464 versus placebo on clinical response as per MMS
Proportion of subjects with symptomatic remission at week 8 | 8 weeks
  To compare the efficacy of ABX464 versus placebo on symptomatic remission
Proportion of subjects with HEMI per Geboes at week 8 | 8 weeks
  To compare the efficacy of ABX464 versus placebo on histologic-endoscopic mucosal

CONTACTS AND LOCATIONS:
Locations (319):
- United States (64):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Lakeview Clinical Research, Guntersville, Alabama
  - GI Alliance, Sun City, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Aurora Care Clinic, Costa Mesa, California
  - Gastro Care Institute, Lancaster, California
  - California Medical Research Associates Inc., Northridge, California
  - Clinnova Research Solutions, Orange, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Clinical Research Of Brandon, LLC, Brandon, Florida
  - Access Research Institute, Brooksville, Florida
  - Auzmer Research, Lakeland, Florida
  - Cfagi, Llc, Maitland, Florida
  - MedOne Clinical Research LLC, Miami, Florida
  - Medical Professional Clinical Research Center, Miami, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida
  - Endoscopic Research, Inc., Orlando, Florida
  - Advanced Research Institute, Inc., Orlando, Florida
  - Gastroenterology Associates of Pensacola, PA, Pensacola, Florida
  - Theia Clinical Research Centers, LLC, Temple Terrace, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - One Health Research Clinic Atlanta, LLC, Norcross, Georgia
  - Eagle Clinical Research, Chicago, Illinois
  - GI Alliance, Glenview, Illinois
  - GI Alliance, Gurnee, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - University of Louisville Research Foundation, Louisville, Kentucky
  - GI Alliance - Baton Rouge, Baton Rouge, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Lucida Clinical Trials LLC, New Bedford, Massachusetts
  - Digestive Health Center PA, Ocean Springs, Mississippi
  - University of Nebraska Medical Center, Omaha, Nebraska
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - Rochester Clinical Research, Rochester, New York
  - Charlotte Gastroenterology and Hepatology, P.L.L.C, Charlotte, North Carolina
  - Care Access Research Lumberton, Lumberton, North Carolina
  - Wilmington Health, Wilmington, North Carolina
  - Gastro Health Research, Cincinnati, Ohio
  - Wexner Medical Center, Columbus, Ohio
  - DSI Research LLC, Springboro, Ohio
  - Columbia Digestive Health Research, Columbia, South Carolina
  - Gastroenterology Associates, PA, Greenville, South Carolina
  - Gastroenterology Center of the MidSouth PC, Germantown, Tennessee
  - GI Alliance - Southlake, Austin, Texas
  - Central Texas Clinical Research, LLC, Austin, Texas
  - Texas Digestive Disease Consultants, Cedar Park, Texas
  - Baylor Scott and White, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - GI Alliance - Garland, Garland, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Biopharma Informatic, Inc. Research Center, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Gastro Health & Nutrition, Katy, Texas
  - GI Alliance - San Marcos, San Marcos, Texas
  - Texas Gastroenterology Associates, Spring, Texas
  - GI Alliance - Webster, Webster, Texas
  - Care Access Research LLC, Ogden, Utah
  - University of Utah, Salt Lake City, Utah
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - TPMG Clinical Research Williamsburg, Williamsburg, Virginia
- Argentina (4):
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes, Buenos Aires
  - STAT Research S.A., Ciudad Autonoma Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Hospital Privado Centro Medico de Cordoba S.A, Córdoba
- Australia (17):
  - Blacktown Hospital, Blacktown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Coral Sea Clinical Research Institute, North Mackay, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Footscray Hospital, Footscray, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Canberra Hospital, Canberra
  - Coral Sea Clinical Research Institute, North Mackay
  - Royal Perth Hospital, Perth
  - Mater Misericordiae Ltd, South Brisbane
- Austria (5):
  - LKH - Universitaetsklinikum Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - KH der Barmherzigen Brüder St.Veit an der Glan, Sankt Veit an der Glan
  - AKH - Medizinische Universität Wien, Vienna
- Belgium (8):
  - AZ Klina, Brasschaat
  - AZ Sint-Lucas, Bruges
  - C. H. U. St-Pierre, Brussels
  - HUB Erasme, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - UZ Leuven, Leuven
  - Clinique CHC MontLégia, Liège
  - CHU UCL Namur, Yvoir
- Bulgaria (5):
  - Medical center Medconsult Pleven OOD, Pleven
  - DCC "Alexandrovska", EOOD, Sofia
  - UMHAT 'Tsaritsa Yoanna - ISUL', EAD, Sofia
  - UMHATEM 'N.I. Pirogov', EAD, Sofia
  - UMHAT Prof. Dr. Stoyan Kirkovich AD, Stara Zagora
- Canada (4):
  - Gastroenterology and Internal Medicine Research Institute, Edmonton, Alberta
  - Scott Shulman Medicine Professional Corporation, North Bay, Ontario
  - Kensington Screening Clinic, Toronto, Ontario
  - McGill University Health Centre- Montreal General Hospital, Montreal, Quebec
- China (51):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Yijishan Hospital of Wannan Medical College, Wuhu, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The 900th Hospital of The Chinese People's Liberation Army Joint Logistics Support Force, Fuzhou, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Yuexiu, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi Zhuang
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi Zhuang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xiangya Hospital, Central South University, Changsha, Hu'nan
  - The 2nd Xiangya Hospital of Central South University, Changsha, Hu'nan
  - The First Affiliated Hospital of University of South China, Hengyang, Hu'nan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - ongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Renmin Hospital, Wuhan University, Wuhan, Hubei
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Jiangxi Gannan Medical College Affiliated 1 st Hospital, Ganzhou, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Taian City Central Hospital, Tai’an, Shandong
  - Ruijin Hospital of Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Renji Hospital Shanghai Jiaotong University School of Medicine - West Branch, Shanghai, Shanghai Municipality
  - Army Specialty Medical Center of The Chinese People's Liberation Army, Chongqing, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Tianjin Union Medical Center, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yun'nan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - West China Hospital, Sichuan University, Sichuan
- Czechia (7):
  - CCR Brno, s.r.o., Brno
  - SurGal Clinic s.r.o., Brno
  - Vojenska nemocnice Brno, Brno
  - Hepato-Gastroenterologie HK s.r.o., Hradec Králové
  - PreventaMed s.r.o., Olomouc
  - CCR Ostrava s.r.o., Ostrava
  - Nemocnice Slany, Slaný
- France (12):
  - CHU Reims - Hôpital Robert Debré, Reims, Ardennes
  - CHU Dijon - Hôpital Bocage Central, Dijon, Cote D'or
  - CHU Besançon - Hôpital Jean Minjoz, Besançon, Doubs
  - CHU Bordeaux - Hôpital Haut-Lévêque, Pessac, Gironde
  - Hopital Saint Eloi, Montpellier, Herault
  - CHU Nantes - Hôtel Dieu, Nantes, Loire Atlantique
  - CHU Saint Etienne - Hôpital Nord, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - CHU Clermont Ferrand - Hopital d'Estaing, Clermont-Ferrand, Puy De Dome
  - Centre Hospitalier de Pau - Hôpital François Mitterrand, Pau, Pyrénées Atlantique
  - Hôpital Henri Mondor, Créteil, Val De Marne
  - Hôpital Bicêtre, Le Kremlin-Bicêtre, Val De Marne
  - Hôpital Saint-Louis, Paris
- Germany (11):
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Praxis fuer Gasroenterologie Prof. Dr. med Robert Ehehalt, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - LMU - Campus Grosshadern, Munich, Bavaria
  - Staedisches Klinikum Brandenburg, Brandenburg, Brandenburg
  - Universitaetsklinikum Frankfurt Goethe-Universitaet, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel, Kiel, Schleswig-Holstein
  - Gastroenterologie Berlin Karlshorst, Berlin
  - Charité - Campus Benjamin Franklin, Berlin
- Greece (5):
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - General Hospital of Athens "Evangelismos", Athens
  - Corfu General Hospital "St. Eirini", Corfu
  - University General Hospital of Heraklion, Heraklion
  - General Hospital of Thessaloniki "Hippokration", Thessaloniki
- Hungary (6):
  - Bekes Varmegyei Kozponti Korhaz, Békéscsaba
  - Clinexpert Kft., Budapest
  - Semmelweis Egyetem, Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Debreceni Egyetem, Debrecen
  - Vas Varmegyei Markusovszky Egyetemi Oktatokorhaz, Szombathely
- India (17):
  - Navneet Memorial Hospital 'Sushrusha', Ahmedabad, Gujarat
  - Shree Giriraj Multispeciality Hospital, Rajkot, Gujarat
  - Unity Hospital ICU and Trauma, Surat, Gujarat
  - Fortis Memorial Research Institute, Gurgaon, Haryana
  - M. S. Ramaiah Medical College and Hospital, Bangalore, Karnataka
  - K.L.E. Society's Dr. Prabhakar Kore Hospital and Medical Research Centre, Belagāve, Karnataka
  - Amrita Institute Of Medical Sciences and Research Centre, Kochi, Kerala
  - King Edward Memorial Hospital Research Centre, Mumbai, Maharashtra
  - Kingsway Hospital, Nagpur, Maharashtra
  - Midas Multispeciality Hospital Pvt Ltd, Nagpur, Maharashtra
  - Chopda Medicare & Research Centre, Nashik, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Sahyadri Specialty Hospital, Pune, Maharashtra
  - Dayanand Medical College and Hospital, Ludhiana, Punjab
  - S. R. Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - Chhatrapati Shahuji Maharaj (CSM) Medical University, Lucknow, Uttar Pradesh
  - Nil Ratan Sircar Medical College, Kolkata, West Bengal
- Italy (13):
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - I.R.C.C.S Policlinico San Donato, San Donato Milanese, Milano
  - Ospedale Sacro Cuore Don Calabria, Negrar, Verona
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Azienda Ospedaliera Giuseppe Brotzu, Cagliari
  - Presidio Ospedaliero Garibaldi Nesima, Catania
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - Ospedale Sacro Cuore Don Calabria, Negrar
  - Azienda Ospedaliera Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisana (Presidio di Cisanello), Pisa
  - Ospedale San Bortolo di Vicenza, Vicenza
- Netherlands (6):
  - Amsterdam UMC, Locatie AMC, Amsterdam
  - Radboud UMC, Nijmegen
  - Erasmus MC, Rotterdam
  - Zuyderland Medisch Centrum - Sittard-Geleen, Sittard
  - ETZ Elisabeth, Tilburg
  - Bernhoven Uden, Uden
- Poland (17):
  - Przychodnia Specjalistyczna Insula, Bełchatów
  - Szpital Zakonu Bonifratow Sp. z o.o., Katowice
  - Centrum Medyczne PROMED, Krakow
  - NZOZ Centrum Medyczne ProMiMed, Krakow
  - AMICARE spółka z ograniczoną odpowiedzialnością spółka komandytowa, Lodz
  - Twoja Przychodnia Opolskie Centrum Medyczne, Opole
  - SOLUMED Centrum Medyczne, Poznan
  - NSZOZ Termedica - Centrum Badan Klinicznych, Poznan
  - Twoja Przychodnia PCM, Poznan
  - Kiepury Clinic MAŁGORZATA JARNOT SPECJALISTYCZNA PRAKTYKA GINEKOLOGICZNO-POŁOŻNICZA, Sosnowiec
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne Sp. z o. o., Szczecin
  - Centrum Zdrowia MDM, Warsaw
  - NZOZ VIVAMED Jadwiga Miecz, Warsaw
  - PlanetMed sp. z o.o., Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
  - ETG Zamosc, Zamość
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej w Lecznej, Łęczna
- Portugal (5):
  - Hospital de Braga, Braga
  - Hospital da Senhora da Oliveira Guimarães, Guimarães
  - Hospital da Luz, Lisbon
  - Centro Hospitalar de Entre o Douro e Vouga, E.P.E - Hospital de São Sebastião, Santa Maria da Feira
  - Centro Hospitalar do Alto Minho - Unidade Local de Saúde do Alto Minho, EPE, Viana do Castelo
- South Korea (20):
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Yeungnam University Hospital, Daegu, Gyeongsangbuk-do
  - Inje University Haeundae Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - The Catholic University of Korea, Daejeon St. Mary's Hospital, Daejeon
  - Gachon University Gil Medical Center, Incheon
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
- Spain (7):
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Clinica Gaias - Santiago, Santiago de Compostela, La Coruña
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Switzerland (4):
  - Claraspital, Basel
  - Inselspital - Universitaetsspital Bern, Bern
  - Intesto Gastroenterologische Praxis, Crohn-Colitis-Zentrum Bern, Bern
  - Universitaetsspital Zuerich, Zurich
- Turkey (Türkiye) (8):
  - Gazi University Medical Faculty, Ankara
  - Koc University Hospital, Istanbul
  - Medicana Kadikoy Hospital, Istanbul
  - Acibadem Kozyatagi Hospital, Istanbul
  - Ege University Medical Faculty, Izmir
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Mersin University Medical Faculty, Mersin
  - Varlik Mah. Kazim Karabekir Cad., Muratpaşa
- Ukraine (15):
  - CNE Cherkasy Regional Hospital of Cherkasy Regional Council, Cherkasy
  - RCNE Chernivtsi Regional Clinical Hospital Gastroenterology Subdivision Bukovinian SMU, Chernivtsi
  - Dnipro Division Medical Center Clinic of Family Medicine of LLC, Dnipro
  - CNE Regional Clinical Hospital of Ivano-Frankivsk Regional Council, Ivano-Frankivsk
  - CNCE Khmelnytskyi Regional Hospital of Khmelnytskyi Regional Council, Khmelnytskyi
  - CNCE Kyiv City Clinical Hospital #1 of Executive Body of Kyiv City Council, Kyiv
  - Clinical Hospital Feofaniia of State Management of Affairs, Kyiv
  - Medical Center of Limited Liability Company Medical Center Concilium Medical, Kyiv
  - Medical Center of Limited Liability Company Saliutas, Lviv
  - CNCE of Lviv Regional Council Lviv Regional Clinical Hospital, Lviv
  - LLC Medical Center The Clinic of Hospodarskyy, Ternopil
  - CNE Uzhhorod city MCH of UCC Dept of Therapy, Uzhhorod
  - Limited Liability Company Medical Center Health Clinic, Medical Clinical Research Center, Vinnytsia
  - CNE M.I. Pyrohov Vinnytsia RCH of Vinnytsia Regional Council, RSC Gastro Center, Vinnytsia
  - Clinic of the SRI of Invalid Rehab (EST Complex) of Pirogov Memorial NMU, Vinnytsia
- United Kingdom (8):
  - Royal London Hospital, London, Greater London
  - King's College Hospital, London, Greater London
  - Hammersmith Hospital, London, Greater London
  - Bury Care Organisation, Bury, Greater Manchester
  - St Mark's Hospital, Harrow, Middlesex
  - Yeovil District Hospital, Yeovil, Somerset
  - Huddersfield Royal Infirmary, Huddersfield, West Yorkshire
  - The Ulster Hospital, Belfast